CLINICAL TRIAL: NCT00220129
Title: Neoadjuvant Epirubicin, Cisplatin and Capecitabine (Xeloda) [ECX] Followed by Definitive Chemoradiation With or Without Surgery for Patients With Newly Diagnosed Localized Squamous Cell Carcinoma of the Oesophagus
Brief Title: Neoadjuvant Epirubicin, Cisplatin and Capecitabine (ECX) Followed by Definitive Chemoradiation With/Without Surgery for Squamous Cell Carcinoma of the Oesophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2186
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Oesophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Epirubicin; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epirubicin, Cisplatin, Capecitabine
Procedure: Surgical Resection

SUMMARY:
This is a study to investigate the efficacy and safety of epirubicin, cisplatin and capecitabine (ECX) as neoadjuvant therapy prior to radical chemoradiotherapy using capecitabine and cisplatin as radio-sensitisers in patients with newly diagnosed localized squamous cell carcinoma of the oesophagus.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histologically verified squamous cell carcinoma of the cervical or thoracic oesophagus
* American Joint Committee on Cancer (AJCC) Stage I-III (T1-3 N0-1 M0) (33), as assessed by spiral or multi-slice computed tomography (CT) and endoscopic ultrasound, where radical chemoradiation would be considered with curative intent.
* No previous chemotherapy, radiotherapy or other investigational drug treatment for this indication.
* World Health Organization (WHO) performance status 0,1 or 2.
* Adequate bone marrow function with platelets > 100 x 10^9/l; white blood cells (WBC) > 3 x 10^9/l; neutrophils > 1.5 x 10^9/l at the time of study entry.
* Serum bilirubin < 35 micromol/l.
* Serum creatinine < 180 micromol/l and measured creatinine clearance over 60 ml/min.
* No concurrent uncontrolled medical condition.
* No previous malignant disease other than non-melanotic skin cancer or carcinoma in situ of the uterine cervix in the last 10 years.
* Life expectancy > 3 months.
* Adequate contraceptive precautions if relevant.
* Informed written consent.

Exclusion Criteria:

* The presence of locally advanced or metastatic disease precluding curative chemoradiation (T4 or Stage IV or M1a-b) or disease not encompassable in a radical radiotherapy field.
* Total dysphagia (O'Rourke's swallowing function scoring system 5) precluding swallowing of capecitabine even when crushed.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Intracerebral metastases or meningeal carcinomatosis.
* New York Heart Association classification Grade III or IV.
* Uncontrolled angina pectoris.
* Pregnancy or breast feeding.
* Impaired renal function with measured creatinine clearance less than 60 ml/min.
* Previous investigational study drug
* Known malabsorption syndromes
* Patients with a known hypersensitivity to fluorouracil (5-FU) or with a dihydropyrimidine dehydrogenase (DPD) deficiency
* Hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-11

PRIMARY OUTCOMES:
2 year overall survival

SECONDARY OUTCOMES:
Objective clinical response rate assessed by computed tomography (CT), endoscopic ultrasound (EUS) and endoscopic biopsy
Pattern of treatment failure
Progression free survival
Proportion of patients not achieving clinical complete response and requiring surgery after chemoradiation
Treatment related toxicity
Time to improvement of dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom